CLINICAL TRIAL: NCT06107296
Title: Early Perioperative Quality Of Recovery After Hip and Knee Arthroplasty: a Retrospective Comparative Cohort Study
Acronym: EARLY-QoR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8898
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Arthroplasty, Hip Replacement; Arthroplasty, Knee Replacement
Keywords: Arthroplasty; Hip Replacement; Knee Replacement; QoR-15 questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hip and knee replacements are indicated to improve long-term quality of life and pain. These long-term results may depend on the quality of the initial postoperative recovery.

However, early postoperative health status after total hip arthroplasty (THA) and total knee arthroplasty (TKA) is not accurately described. Through this retrospective study, the investigators wanted to describe the perioperative state of health monitored using the QoR-15 questionnaire for THA and TKA patients from the perioperative moment to postoperative day 28.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years)
* Having benefited from an ATG or ATH at Strasbourg University Hospital between March 1, 2020 and December 31, 2022
* Tracked with QoR-15 score
* Patient not opposing the reuse of his data for scientific research purposes

Exclusion Criteria:

* Refusal to participate in the study
* Patient admitted to THA for a hip fracture
* Patient admitted for multiple THA or TKA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (age ≥ 18 years) Having benefited from an ATG or ATH at Strasbourg University Hospital between March 1, 2020 and December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Mean QoR-15 score at the preoperative period and postoperative days 1, 3, 14 and 28 | At the preoperative period and postoperative days 1, 3, 14 and 28
  Perioperative health status monitored using the QoR-15 questionnaire for THA and TKA patients from perioperative time to postoperative day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésiologie - Réanimation Chirurgicale - CHU de Strasbourg - France, Strasbourg, France